CLINICAL TRIAL: NCT05673798
Title: Development and Validation of Nomogram Predicting Survival in Chinese SCLC Patients
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: ChineseSCLC2022
Record Dates: First submitted 2022-11-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- training cohort: The investigators used the training cohort to develop the predictive nomogram with potential risk factors( initial response to chemotherapy)
  Interventions: Other: initial chemotherapy response
- validation cohort: The investigators used the validation cohort to verify the clinical utility and predictive ability
  Interventions: Other: initial chemotherapy response

INTERVENTIONS:
Other: initial chemotherapy response — Initial chemotherapy response is the first imaging examination of SCLC patient after starting chemotherapy

SUMMARY:
In this retrospective study, patients diagnosed with SCLC between January 2011 to September 2022 were identified from database of the Second Hospital of Shandong University. Following inclusion criteria should be met: (1) Had histologically or cytologically confirmed newly diagnosed SCLC; (2) No cancer treatment has been done before; (3) Complete clinical, laboratory, imaging, treatment data and follow-up information. The exclusion criteria included: Patients without complete records for pathological information, complete epidemiology and other key clinical information.

DETAILED DESCRIPTION:
The investigators classified qualitative variables according to clinical practice. Age included less than 60 years, 61-66 years, and more than 67 years. The primary tumor location included left-sided and right-sided. The anatomic sites included lower and others. The smoking status included never smoker and ever smoker. The forms of performance status according to the Eastern Cooperative Oncology Group scale (ECOG PS) were ECOG ≤ 2, and ECOG ≥ 3. Five groups were formed according to clinical T stage (T0-1, T2, T3, T4, and T stage that could not be evaluated). Three groups were formed according to clinical N stage (N0-1, N2-3, and N stage that could not be evaluated). Some stages were unevaluated, on account of a portion of non-measurable tumor size and lymph node. Three groups were formed according to clinical M stage (M0, Ma-b, Mc). Four groups were formed according to clinical TNM stage (Ⅰ-Ⅱ, Ⅲ, Ⅳ and TNM stage that could not be evaluated). The common metastatic sites(brain, liver, and bone) of tumor was divided into none and yes. The hematologic markers (serum natrium , lactate dehydrogenase, carcinoembryonic antigen, neuron-specific enolase, cytokeratin 19 fragment, and pro-gastrin-releasing peptide) were divided into normal and abnormal. The above information was collected before treatment. The RECIST version 1.0 was used to assess tumor responses after initial imaging studies of commencing chemotherapy. Initial chemotherapy response is the first imaging examination of SCLC patient after starting chemotherapy. Six groups were formed according to initial response to chemotherapy (CR, PR, SD, PD, response that could not be evaluated, and no chemotherapy). Other treatments (radiotherapy, surgery, targeted therapy, immunotherapy, Interventional therapy, and whole-brain prophylactic cranial irradiation) was classified none and yes.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosis of small cell lung cancer
2. No cancer treatment has been done before
3. Complete clinical, laboratory, imaging, treatment data and follow-up information

Exclusion Criteria:

1. Without complete records for pathological information, complete epidemiology and other key clinical information

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In this retrospective study, patients diagnosed with SCLC between January 2011 to September 2022 were identified from database of the Second Hospital of Shandong University.
Sampling Method: Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival | January 2011 to September 2022
  the Time Between the Discovery of the Tumor and the Patient's Death

REFERENCES:
- [Background] Lara PN Jr, Redman MW, Kelly K, Edelman MJ, Williamson SK, Crowley JJ, Gandara DR; Southwest Oncology Group. Disease control rate at 8 weeks predicts clinical benefit in advanced non-small-cell lung cancer: results from Southwest Oncology Group randomized trials. J Clin Oncol. 2008 Jan 20;26(3):463-7. doi: 10.1200/JCO.2007.13.0344. PMID 18202421